CLINICAL TRIAL: NCT01825122
Title: Efficacy and Safety of Βeta-adrenoceptor Inverse Agonist and Biased Ligand, Nadolol, In Smoking Cessation of Patients With Chronic Cough With or Without Airflow Obstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Invion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INVSC001
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nadolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Active, nadolol (Experimental): Active
  Interventions: Drug: Nadolol

INTERVENTIONS:
Drug: Nadolol
  Arms: Active, nadolol
Drug: Placebo
  Arms: Placebo

SUMMARY:
To test the hypothesis that treatment with the inverse agonist nadolol will improve smoking cessation in patients with chronic cough associated with long-term smoking, with or without airflow obstruction, including those with established chronic obstructive pulmonary disease (COPD) (chronic bronchitis dominant) or non-obstructive chronic bronchitis (NCB), compared to placebo and standard of care, while undergoing a validated smoking cessation program.

ELIGIBILITY:
Inclusion Criteria:

Potential study participants will be referred from approved smoking cessation programs or be willing to enter a smoking cessation program administered by the participating sites. Individuals who meet all of the following criteria at Visit 1 are eligible for enrollment as study participants:

1. Active cigarette-smoking males and females between the ages of 18-70 with chronic cough associated with long-term smoking, with or without airflow obstruction, including Non-obstructive chronic bronchitis (NCB) or physician-diagnosed COPD (chronic bronchitis dominant), as defined by the American Thoracic Society.
2. Committed desire to quit smoking in conjunction with participation in an approved smoking cessation program administered by the participating sites. Enrollment in the smoking cessation program must take place prior to Visit 3 (third dose escalation visit).
3. Diagnosis of COPD (chronic bronchitis dominant) or NCB, or presenting with chronic cough associated with long-term smoking.
4. Pre-bronchodilator FEV1 greater than 55% of predicted
5. Baseline blood pressure ≥ 110/65mm Hg
6. Baseline heart rate ≥ 60 beats/min.
7. Smoking at least 10 cigarettes per day prior to participation in the approved smoking cessation program.
8. Self-reported prior failure(s) to quit smoking during participation in a smoking cessation program.
9. Able to complete diary cards and comply with study procedures.
10. Females of childbearing age may participate only if they have a negative pregnancy test, are non-lactating, and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study.

Exclusion Criteria:

Subjects who meet ANY of the following criteria are not eligible for enrollment:

1. Diagnosis of asthma, cystic fibrosis, or PiZZ emphysema
2. Inability or unwillingness to give written informed consent
3. History of upper/lower respiratory tract infection, COPD exacerbation requiring systemic steroids, antibiotics, and or ER visit or urgent care within 6 weeks of Visit 1
4. History of adverse reaction or allergy to nadolol
5. History of neurological, hepatic, renal, or other medical conditions that may interfere with the interpretation of data or the patient's participation in the study or may increase safety concerns
6. History of cardiovascular diseases including uncontrolled hypertension (BP >160/100), ischemic heart disease, congestive heart failure (NYHA III or IV), valvular heart disease or cardiomyopathy
7. Known allergy or sensitivity to atropine or ipratropium bromide
8. Documented or self-reported current history of alcoholism or drug abuse
9. Participation in another research trial within 30 days of starting this trial
10. Unwillingness or inability to comply with study procedures
11. Inability to swallow the study medication
12. Pregnant or nursing
13. Current use of any OTC remedies containing pseudoephedrine, ephedrine-based or containing dietary or herbal supplements.
14. Scheduled for surgery requiring general anaesthesia
15. Referred for smoking cessation without serious commitment to quit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Castro, M.D., Principal Investigator — Washington University of St. Louis
Locations (4):
- United States (4):
  - Hope Research Center, Phoenix, Arizona
  - Nuren Medical, Miami, Florida
  - Abel Buchheim Pharmaceutical Research, Miami, Florida
  - Washington University School of Medicine, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- Active, Nadolol: Active
  Nadolol
Period: Overall Study
Arm/Group | Placebo | Active, Nadolol
Started | 77 | 78
Completed | 67 | 59
Not Completed | 10 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active, Nadolol | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 76 | 143
  >=65 years | 10 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.08 (13.58) | 44.08 (12.52) | 46.06 (13.17)
Gender [Count of Participants; unit: Participants]
  Female | 45 | 33 | 78
  Male | 32 | 45 | 77
Region of Enrollment [Number; unit: participants]
  United States | 77 | 78 | 155

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Number of Cigarettes Smoked Per Day
Time Frame: Baseline to end of treatment, up to 15 weeks
Population: The analysis population reflects all patients who achieved maintenance dosing, including those who did not complete the study
Measure: Number; unit: participants
Arm/Group | Placebo | Active, Nadolol
Number analyzed (Participants) | 72 | 73
participants
  ≥ 70% Reduction from Baseline | 36 | 45
  < 70% reduction from baseline | 36 | 28

ADVERSE EVENTS:
Time Frame: Up to 30 days following discontinuation of the study, for up to 21 weeks
Arm/Group | Placebo | Active, Nadolol
Serious Adverse Events (participants affected / at risk) | 1/77 | 2/78
Other Adverse Events (participants affected / at risk) | 34/77 | 35/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=77) | Active, Nadolol (N=78)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bipolar episode (Psychiatric disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | Active, Nadolol (N=78)
Dizziness (Cardiac disorders) | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Dry mouth (Gastrointestinal disorders) | 17 | 21
Dysgeusia (Gastrointestinal disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less